CLINICAL TRIAL: NCT03304665
Title: Recruitment and Characterization of Healthy Research Volunteers for NIMH Intramural Studies
Status: Recruiting | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170181; 17-M-0181
Record Dates: First submitted 2017-10-06; First posted 2017-10-09 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08-22

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; Mental Health; Common Data Elements
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Healthy Volunteers

SUMMARY:
Objective: To screen and create a list of adult volunteers in good health for participation in research studies conducted at the National Institutes of Health (NIH) in Bethesda, Maryland. Develop a normative set of structural and functional brain MRI scans that are linked to healthy research volunteer characteristics. Maximize scientific impact of data from volunteers by broadly sharing with other researchers.

Study Population: Adult males and females in general good health who are 18 years of age and older.

Design: Adult individuals who are interested in participating in NIMH IRP clinical studies as a healthy research volunteer can directly visit or be directed to visit the study website where they will first consent electronically and then complete a set of online self-report measures. Items may include: demographic information, mental health symptoms, disability status, substance use patterns, handedness and clinical/family history. Individuals who are flagged based on predetermined responses to survey items will be further screened by a member of the study clinical team. If found to be ineligible for the study because of a clinically significant or unstable medical or mental health condition, these individuals will be referred back to the community and/or given information about NIMH clinical studies for which they may be eligible. Respondents with no flags or who pass through additional screening will be scheduled for an in-person assessment. During the outpatient appointment and after in-person informed consent, participants will receive a brief clinical interview to screen for current medical and mental conditions, and risk for self-harm. They will complete assessments of psychological, emotional, physiologic, biological and cognitive functioning. Participants will undergo a physical exam and be asked to provide blood and urine samples for routine clinical labs. Participants can separately consent for an optional baseline brain magnetic resonance imaging (MRI) scan and an optional magnetoencephalography (MEG) exam. All consent forms will explicitly inform participants that if enrolled in the study, their de-identified data will be broadly and publicly shared through NIH-approved data repositories. Participants in this recruitment and characterization study will then be placed on a list of healthy research volunteers from which other NIMH IRP studies may recruit according to the inclusion and exclusion criteria in their respective IRB-approved protocols.

Outcome Measures: Outcome measures may include demographic data, mental and medical history and symptoms, results of psychological, emotional, physiologic, biological, and cognitive testing, physical exam and MRI findings....

DETAILED DESCRIPTION:
Objective: To screen and create a list of adult volunteers in good health for participation in research studies conducted at the National Institute of Mental Health (NIMH) in Bethesda, Maryland. Develop a normative set of structural and functional brain MRI scans and MEG recordings that are linked to healthy research volunteer characteristics. Maximize scientific impact of data from volunteers by broadly sharing with other researchers.

Study Population: Adult males and females in general good health who are 18 to 70 years of age.

Design:

This study has 2 parts. Part 1 is an online screen in which interested participants are asked to complete online forms that will help determine their eligibility for Part 2, which is an in-person assessment at the NIH Clinical Center. In addition, there are 3 optional procedures, an optional MRI brain scan, MEG recording, and electrocardiography (EKG) that are completed at the NIH Clinical Center. Procedures are done in sequence unless a person is found to be ineligible to move to the next step.

Adult individuals who are interested in participating in NIMH IRP clinical studies as a healthy research volunteer can directly visit or be directed to visit the study website where they will first consent electronically and then complete a set of online self-report measures. Items may include: demographic information, mental health symptoms, psychological measures, disability status, substance use patterns, and clinical/family history. Individuals who are flagged based on predetermined responses to survey items may be further screened by a member of the study clinical team. If found to be ineligible for the study because of a clinically significant or unstable medical or mental health condition, these individuals will be referred back to the community and/or given information about NIMH clinical studies for which they may be eligible. Respondents with no flags or who pass through additional screening will be eligible for a clinical (in-person) assessment at the NIH Clinical Center. During the in-person outpatient appointment the participant will provide informed consent for the clinical assessment and optional MRI and MEG studies. At that point they are considered enrolled in the study. The clinical assessment may include safety assessment, vital signs, history and physical, labs, cognitive tests, mental health surveys, and structured psychiatric diagnostic interview.

Some assessments may be conducted either in-person or virtually using approved telehealth services. Laboratory tests will be done for routine clinical purposes. The consent form will explicitly inform participants that if enrolled in the study, their de-identified data will be broadly and publicly shared through NIH-approved data repositories. Participants in this recruitment and characterization study may then be placed on a list of healthy research volunteers and their contact information may be shared with other NIMH IRP studies.

Outcome Measures:

* Primary outcome measure - List of well characterized healthy volunteers including demographic, psychological, physical, laboratory, MEG, and MRI data; and utilization of volunteer participants by NIMH IRP investigators.
* Secondary outcome measure - Upload of de-identified healthy volunteer characterization data to an open access data repository for secondary research purposes; data may include demographic, psychological, physical, laboratory, MEG, and MRI measures.

ELIGIBILITY:
* INCLUSION CRITERIA:
* 18 - 70 years of age.
* Able to read, speak, and understand English.
* Able to provide informed consent.
* In current good general health.

EXCLUSION CRITERIA:

* Have a history of significant or unstable medical or mental health condition requiring treatment, such as heart or lung disease, depression or psychosis.
* Endorse current self-injury, suicidal thoughts or behavior.
* Have current illicit drug use by history or urine drug screen.
* Are found to have an abnormal physical exam or laboratory result that may require treatment or further evaluation.
* Less than an 8th grade education.
* Pregnancy.
* Positive HIV test as HIV positivity has been associated with neurological changes.

Optional Brain MRI scan exclusion criteria:

* Metal in body which would make having an MRI scan unsafe.
* Being uncomfortable in small, closed spaces such as the MRI machine.
* Inability to lie comfortably on back for at least 45 minutes.
* Pregnancy.

Optional MEG recording exclusion criteria:

-Metal in body which would cause artifacts on MEG recordings.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy research volunteers
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2027-04-26 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Online self-report and in-person assessments that may yield demographic data, mental and medical history and symptoms, results of measures of psychological, emotional, physiologic, biological, and cognitive functioning, and physical or MRI findi... | Ongoing
  Online self-report and in-person assessments that may yield demographic data, mental and medical history and symptoms, results of measures of psychological, emotional, physiologic, biological, and cognitive functioning, and physical or MRI findings.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Zarate, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-M-0181.html